CLINICAL TRIAL: NCT04061915
Title: HIV Oral Testing Infographic Experiment (HOTIE)
Brief Title: HIV Oral Testing Infographic Experiment
Acronym: HOTIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018-1573; R25MH087217 (NIH); P30MH062294 (NIH)
Record Dates: First submitted 2019-07-17; First posted 2019-08-20 (Actual); Results first posted 2022-03-23 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-03

CONDITIONS: HIV/AIDS
Keywords: HIV Prevention; Sexual and Gender Minorities; Consumer Health Informatics
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Coitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infographic Intervention (Experimental): Participants in the intervention arm will view an HIV self-testing infographic.
  Interventions: Behavioral: Infographic Intervention
- Control (Active Comparator): Participants in the control arm will read paper-based HIV self-testing instructions.
  Interventions: Behavioral: Paper-based HIV self-testing information

INTERVENTIONS:
Behavioral: Infographic Intervention — The intervention consists of participants viewing an HIV self-testing infographic.
  Arms: Infographic Intervention
Behavioral: Paper-based HIV self-testing information — The control arm will read paper-based HIV self-testing instructions.
  Arms: Control

SUMMARY:
Premised on the National AIDS Strategy's focus on identifying new HIV infections through increased HIV testing, the purpose of this formative pilot study is to develop and test an integrated HIV self-testing strategy that utilizes a simplicity-model approach to HIV self-testing in emerging adult sexual minority men of color.

DETAILED DESCRIPTION:
In the United States, approximately 1.1 million persons are living with HIV. Despite novel pharmacological breakthroughs, comprehensive models of health care, and targeted HIV testing initiatives, over 160,000 persons are still unaware of their HIV serostatus. Emerging adult, sexual minority, men of color are disproportionately affected. Premised on the National AIDS Strategy's focus on identifying new HIV infections through increased HIV testing, the purpose of this formative pilot study is to develop and test an integrated HIV self-testing strategy that utilizes a simplicity-model approach to HIV self-testing in emerging adult sexual minority men of color.

The overall study will focus on: (a) understanding facilitators and barriers to HIV self-testing among emerging adult MSM, (b) designing a HIV self-testing infographic that utilizes a simplicity model, (c) finalizing the HIV self-testing infographic with input from a leadership group of HIV community members, (d) conducting a pilot clinical trial with 300 emerging adult (ages 18-34), sexual minority, men of color to test if a collaboratively-designed HIV self-testing infographic can facilitate accurate and effective understanding of how to self-test for HIV when compared to paper-based, HIV self-testing information.

By conducting this study, we will gain beneficial insights necessary for presenting HIV self-testing instructions in a meaningful, relevant, and comprehensible way. The results of this pilot study have the potential to inform strategies regarding how self-testing instructions can be worded or visually presented in order to break both literacy and language barriers that affect testing utilization and results accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Understand and read English
* Assigned male sex at birth
* Self-identify as gay, same-gender-loving, or MSM
* Self-report being HIV-negative or unknown HIV serostatus

Exclusion Criteria:

• Persons with a known HIV diagnosis

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-reported assigned male sex at birth.
Enrollment: 322 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. Raquel Ramos, PhD, MBA, MSN, FNP-BC, Principal Investigator — New York University Rory Meyers College of Nursing
Locations (1):
- New York University Rory Meyers College of Nursing, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ramos SR, Lardier DT Jr, Bond KT, Boyd DT, O'Hare OM, Nelson LE, Guthrie BJ, Kershaw T. Participatory Design of a Web-Based HIV Oral Self-Testing Infographic Experiment (HOTIE) for Emerging Adult Sexual Minority Men of Color: A Mixed Methods Randomized Control Trial. Int J Environ Res Public Health. 2021 Nov 12;18(22):11881. doi: 10.3390/ijerph182211881. PMID 34831644
- [Derived] Ramos SR, Reynolds H, Johnson C, Melkus G, Kershaw T, Thayer JF, Vorderstrasse A. Perceptions of HIV-Related Comorbidities and Usability of a Virtual Environment for Cardiovascular Disease Prevention Education in Sexual Minority Men With HIV: Formative Phases of a Pilot Randomized Controlled Trial. J Med Internet Res. 2024 Aug 22;26:e57351. doi: 10.2196/57351. PMID 38924481
- [Derived] Ramos SR, Lardier DT Jr, Opara I, Turpin RE, Boyd DT, Gutierrez JI Jr, Williams CN, Nelson LE, Kershaw T. Intersectional Effects of Sexual Orientation Concealment, Internalized Homophobia, and Gender Expression on Sexual Identity and HIV Risk Among Sexual Minority Men of Color: A Path Analysis. J Assoc Nurses AIDS Care. 2021 Jul-Aug 01;32(4):495-511. doi: 10.1097/JNC.0000000000000274. PMID 34101701
- [Derived] Ramos SR, Lardier DT Jr, Boyd DT, Gutierrez JI Jr, Carasso E, Houng D, Kershaw T. Profiles of HIV Risk, Sexual Power, and Decision-Making among Sexual Minority Men of Color Who Engage in Transactional Sex: A Latent Profile Analysis. Int J Environ Res Public Health. 2021 May 7;18(9):4961. doi: 10.3390/ijerph18094961. PMID 34066948
- [Derived] Ramos SR, Lardier DT Jr, Warren RC, Cherian M, Siddiqui S, Kershaw T. Substance Use, General Health and Health Literacy as Predictors of Oral Health in Emerging Adult Sexual Minority Men of Color: A Secondary Data Analysis. Int J Environ Res Public Health. 2021 Feb 18;18(4):1987. doi: 10.3390/ijerph18041987. PMID 33670796

RESULTS

PARTICIPANT FLOW:
Groups:
- Infographic Intervention: Participants randomized to the online intervention arm will review the HIV self-testing infographic. Once reviewed, participants will answer comprehension and preference questions about the self-testing infographic.
  Infographic Intervention: A HIV self-testing infographic that utilizes a simplicity model of pictures with limited text.
- Control: Participants randomized to the control arm will text-based HIV self-testing instructions.
  Text-based HIV self-testing information: The online control arm will consist of text-based, HIV self-testing information.
Period: Overall Study
Arm/Group | Infographic Intervention | Control
Started | 161 | 161
Completed | 161 | 161
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infographic Intervention | Control | Total
Number analyzed (Participants) | 161 | 161 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (4.74) | 26.4 (4.5) | 26.35 (4.66)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male Participants | 161 | 161 | 322
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 79 | 78 | 157
  Not Hispanic or Latino | 82 | 83 | 165
  Unknown or Not Reported | 0 | 0 | 0
HIV Knowledge [Mean (Standard Deviation); unit: units on a scale] — 18-item dichotomous response (true/false) measure that detects an individual's knowledge about HIV transmission, prevention, and consequences. Range = 0 to 18 (higher score indicates higher HIV knowledge)
  units on a scale | 11.29 (4.94) | 11.74 (4.58) | 11.51 (4.76)

OUTCOME MEASURES:

1. Primary Outcome: HIV Self-testing Knowledge
Description: Self-report comprehension questionnaire based on accurate completion of HIV-self testing steps. Measure of participants understanding of the text and pictures on how to perform an HIV self-test.
  Questions asked about using the test stick, oral swabbing, what to do with the test stick after swabbing, minutes of wait time before interpretation of result, comprehension of result. Range: 0 to 5 (5 indicates all correct responses)
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Infographic Intervention: Emerging adults randomized to the online intervention arm will review the self-testing infographic. Once participants finish reviewing, they will answer comprehension and preference questions about the self-testing infographic.
  Infographic Intervention: A HIV self-testing infographic that utilizes a simplicity model collaboratively designed by a leadership group of HIV community members
- Control: Emerging adults randomized to the online control arm will read paper-based HIV self-testing information.
  Paper-based HIV self-testing information: The online control arm will consist of paper-based, HIV self-testing information that the emerging adults will read.
Arm/Group | Infographic Intervention | Control
Number analyzed (Participants) | 161 | 161
score on a scale | 3.24 (1.16) | 3.79 (1.26)

2. Primary Outcome: Usefulness, Ease of Use, Ease of Learning and Satisfaction of the HIV Self-testing Infographic
Description: USE Questionnaire: Usefulness, Satisfaction, and Ease Measures the subjective usability of the HIV self-testing infographic. We used 14-items, using a 7-point Likert, and the minimum score is 14 and maximum 98 to examine dimensions of usability: usefulness, ease of use, ease of learning, and satisfaction. Scores for each dimension are averaged together to get a composite score.We report the overall usability of the infographic.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infographic Intervention
Number analyzed (Participants) | 161
score on a scale | 76.47 (16.62)

3. Secondary Outcome: Health Literacy
Description: Standard Assessment Health Literacy - English (SAHL-E). 18 test items designed to assess an English-speaking adult's ability to read and understand common medical terms. The test could help health professionals estimate the adult's health literacy level. Range - 0 to 18 (Higher score is higher health literacy)
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infographic Intervention | Control
Number analyzed (Participants) | 161 | 161
score on a scale | 15.9 (2.96) | 14.9 (3.98)

ADVERSE EVENTS:
Time Frame: Data collection took place over 6 months. For each participant, adverse event data were collected over the duration of 1 day, which was the amount of total time a participant completed all measures.
Description: This was an online pilot RCT to test the feasibility, acceptability, and comprehension of an HIV self-testing infographic. The risk of serious adverse events, all-cause mortality, and other adverse risks associated with this study was low.
Arm/Group | Infographic Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/161
Serious Adverse Events (participants affected / at risk) | 0/161 | 0/161
Other Adverse Events (participants affected / at risk) | 0/161 | 0/161

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT04061915/Prot_SAP_000.pdf